CLINICAL TRIAL: NCT01109082
Title: Gait and Postural Stability Assessment in Children With Idiopathic Scoliosis Undergoing Posterior Spine Instrumentation
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: DePuy Spine (Industry)
Responsible Party: Principal Investigator, Sahar Hassani, Research Administrator, Shriners Hospitals for Children
Other Study IDs: AIS-2010
Record Dates: First submitted 2010-04-15; First posted 2010-04-22 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Scoliosis
Keywords: Scoliosis; gait; posture; balance
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adolescents with idiopathic scoliosis: Adolescents with idiopathic scoliosis
  Interventions: Procedure: posterior spine fusion

INTERVENTIONS:
Procedure: posterior spine fusion — vertebrae are fused to straighten a spinal curve

SUMMARY:
The goal of this study is to evaluate children and adolescents with idiopathic scoliosis who are undergoing spinal fusion using motion analysis, balance, and outcome questionnaires. Little research has been done to evaluate how different fusion levels impact walking patterns, range of motion, posture and balance following spine instrumentation in children with idiopathic scoliosis. Debate still continues whether posterior spinal instrumentation with the last instrumented vertebra at or above Lumbar 3 (L3) will provide sufficient spine correction, greater motion, and better posture and balance when compared to a child with instrumentation at Lumbar 4 (L4). Furthermore, how does the spine fusion endpoint (last instrumented vertebra) impact quality of life, participation, and impairment in children and adolescents with idiopathic scoliosis and how do they compare to healthy age-matched peers. The goal of this study is to compare these two end points using gait analysis, postural stability, and outcome tools with the hopes of providing better clinical care to children with idiopathic scoliosis.

DETAILED DESCRIPTION:
The study population will include sixty (60) children with idiopathic scoliosis who will undergo spine surgery and sixty (60) developing children "Control Group". Scoliosis patients will undergo a period of testing which requires three visits: pre-operative evaluation, one-year post-operative evaluation, and two-year post-operative evaluation. The Control Group will require one initial assessment. A total of 240 evaluations will be performed over a three-year period. We will evaluate the correlation among outcome tools and quantitative measures in order to determine how these instruments can be used more effectively for better treatment. Subjects and their parents will be fully informed of the nature of the study as well as the potential risk involved and sign the appropriate consent form. The study will be reviewed by the IRB and include HIPAA compliance. This will be accomplished during testing at the Shriners Hospital for Children- Chicago Motion Analysis Lab. All possible steps will be taken to assure the safety and convenience of the study participants. All subjects will be evaluated using clinical outcome tools (PODCI, SF-36) and will undergo quantitative 3-D motion analysis and postural stability assessment. Quantitative 3-D gait analysis will be done with our 14-camera Motion Capture system and passive reflective markers (Figure 3). Motion analysis will be performed with each subject walking at a comfortable and natural speed on the laboratory walkway. Passive markers will be attached to anatomic landmarks in standardized locations using double-backed tape. Marker coordinate data will be used to determine range of motion and joint angles.

Four forceplates will be used to measure kinetic data and static balance. Postural stability testing will be performed on all subjects (Figure 4). We will evaluate responses to dynamic stability challenges that investigates motor and sensory control and adaptation to perturbations. Static (quiet standing) postural stability tests will be done on all subjects. A licensed physical therapist (PT) will perform the exam following the protocol of the Shriners Hospital for Children's motion lab.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic scoliosis
* between the ages of 10 - 20
* need a spine fusion at L4 or above
* can walk on your own
* have not had surgery on spine before

Exclusion Criteria:

* pregnant

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with idiopathic scoliosis that have a Cobb angle greater than 50 degrees.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2007-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Motion Analysis | Pre-Operation visit (within 1 week prior to surgical date)
  Gait and standing spine range of motion are measured using a 3-D motion capture system.
Motion Analysis | 1 Year Post-Operative
  Gait and standing spine range of motion are measured using a 3-D motion capture system.
Motion Analysis | 2 Years Post-Operative
  Gait and standing spine range of motion are measured using a 3-D motion capture system.

SECONDARY OUTCOMES:
Functional Questionnaires | Collected at Pre-Operative visit (1 week prior to surgical date)
  A functional outcome questionnaire filled out by the parents and patient.
Functional Questionnaires | Collected at 1 year post-operative visit
  A functional outcome questionnaire filled out by the parents and patient.
e-med plantar pressures | Collected at Pre-Operative visit (1 week prior to surgical visit)
  A pressure map of the plantar surface of the foot during walking.
Postural Stability | Pre-Operative (1 week prior to surgical visit)
  Standing balance and postural stability are measured using a NeuroCom Equitest System and Twin Forceplate system.
Functional Questionnaires | Collected at 2 year follow up
  A functional outcome questionnaire filled out by the parents and patient.
e-med plantar pressures | Collected at 1 year follow up
  A pressure map of the plantar surface of the foot during walking.
e-med plantar pressure | 2 year follow up
  A pressure map of the plantar surface of the foot during walking.
Postural Stability | 1 Year post-operative visit
  Standing balance and postural stability are measured using a NeuroCom Equitest System and Twin Forceplate system.
Postural Stability | 2 year post-operative follow up
  Standing balance and postural stability are measured using a NeuroCom Equitest System and Twin Forceplate system.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Hassani, MS, Principal Investigator — Shriners Hosptials for Children
Locations (1):
- Shriners Hospitals for Children, Chicago, Illinois, United States